CLINICAL TRIAL: NCT01420549
Title: Phase III, Multicenter, Randomized, Open-label, Comparative Study to Evaluate Efficacy and Safety of Rosuvastatin + Ezetimibe Versus Simvastatin + Ezetimibe in High Risk Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia
Brief Title: Efficacy/Safety of Rosuvastatin+Ezetimibe in High Risk Patients With Primary Hypercholesterolemia/Mixed Dyslipidemia
Acronym: LANCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-TRZ-03(06/11)
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Hypercholesterolemia; Dyslipidemia
Keywords: Hypercholesterolemia; Dyslipidemia
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — Rosuvastatin Calcium; Ezetimibe; Simvastatin; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin + Ezetimibe (Experimental): Participants received Rosuvastatin 10 mg+ Ezetimibe 10 mg tablet orally once daily for 5 weeks and after a LDL evaluation if it level was <100 mg/dL the dose was maintained for more 4 weeks. However, if the LDL-C levels was ≥100 mg/dL, the dose was adjusted to Rosuvastatin 20 mg+ Ezetimibe 10mg tablet orally once daily for more 4 weeks.
  Interventions: Drug: Rosuvastatin 10 mg + Ezetimibe 10 mg and Rosuvastatin 20 mg + Ezetimibe 10 mg, according to clinical evaluation.
- Simvastatin + Ezetimibe (Active Comparator): Participants received Simvastatin 20 mg+ Ezetimibe 10 mg tablet orally once daily for 5 weeks and after a LDL evaluation if it level was <100 mg/dL the dose was maintained for more 4 weeks. However, if the LDL-C levels was ≥100 mg/dL, the dose was adjusted to Simvastatin 40 mg + Ezetimibe 10mg tablet orally once daily for more 4 weeks.
  Interventions: Drug: Simvastatin 20 mg + Ezetimibe 10 mg and Simvastatin 40 mg + Ezetimibe 10 mg, according to clinical evaluation.

INTERVENTIONS:
Drug: Rosuvastatin 10 mg + Ezetimibe 10 mg and Rosuvastatin 20 mg + Ezetimibe 10 mg, according to clinical evaluation. — Tables containing: Rosuvastatin 10 mg + Ezetimibe 10 mg and Rosuvastatin 20 mg + Ezetimibe 10 mg, according to clinical evaluation.
  Other Names: Lance
  Arms: Rosuvastatin + Ezetimibe
Drug: Simvastatin 20 mg + Ezetimibe 10 mg and Simvastatin 40 mg + Ezetimibe 10 mg, according to clinical evaluation. — Tables containing: Simvastatin 20 mg + Ezetimibe 10 mg and Simvastatin 40 mg + Ezetimibe 10 mg, according to clinical evaluation.
  Other Names: Vytorin
  Arms: Simvastatin + Ezetimibe

SUMMARY:
The purpose of this study is to determine the non-inferiority between two different FDC (fixed-dose combination), measuring LDL-Cholesterol levels, in high risk patients with primary hypercholesterolemia or mixed dyslipidemia.

DETAILED DESCRIPTION:
The primary efficacy variable was the percentage of LDL-C variation at the end of nine weeks of treatment, compared to baseline (pre-randomization), in participants who achieved LDL <100 mg/dL were considered to have been successfully treated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 to 80 years;
* Participants diagnosed with primary hypercholesterolemia or mixed dyslipidemia;
* Participants must not have other clinically significant comorbidities that may interfere with study evaluations;
* Participants able to understand and adhere to the therapeutic scheme and to attend the study visits;
* Participants who agree to maintain a low cholesterol diet throughout the study;
* Participants who agree to discontinue previous medication for hypercholesterolemia treatment throughout the study;
* Participants with hypercholesterolemia or mixed dyslipidemia with the following laboratory test results on the baseline visit: LDL-C level >130 mg/dl if were receiving prior treatment with statins; or LDL-C level >100 mg/dl if were receiving prior treatment with first generation statins; or LDL ≥160 mg/dL and ≤220 mg/dL and triglycerides ≤350 mg/dL if were not in prior treatment with statins.
* Female participants in reproductive age with negative serum beta-hCG test result in the baseline visit who agree to use acceptable contraceptive methods (oral contraceptives, injectable contraceptives, intrauterine device (IUD), hormonal implants, barrier methods, hormonal patch, tubal ligation or female participants who declare to perform non reproductive sexual practices); except surgically sterile (for example oophorectomy and hysterectomy), surgical sterilization or of the partner; or postmenopausal for at least one year;
* Participants with laboratorial test results after treatment with Simvastatin 20 mg for four weeks with LDL-C level ≥100 mg/dl.

Exclusion Criteria:

* Heart failure class III or IV (NYHA- New York Heart Association);
* Blood dyscrasia;
* Unstable angina pectoris;
* Myocardial infarction in the last 3 months;
* Planning for CABG (coronary artery bypass graft), peripheral or carotid percutaneous intervention for the next 90 days;
* Renal insufficiency: estimated Glomerular Filtration Rate (GFR) < 30 ml/min/m2;
* History of alcoholism that, at the investigator's discretion, could compromise the drug treatment compliance;
* Participants with comorbidities that hinder the interpretation of results or contraindicate the lipid-lowering therapy [uncontrolled hypothyroidism (thyroid-stimulating hormone [TSH] > 8 mUI/mL); uncontrolled diabetes (Hemoglobin A1c [HbA1c] > 8%); active hepatic disease; antiretroviral therapy for HIV, neoplasm (except for adequately treated skin cancer within the past 5 years), concomitant immunosuppressive therapy (transplant receivers and rheumatic disease);
* Uncontrolled systemic arterial hypertension;
* Hypersensitivity to any component of the investigational product;
* Participant who has participated in clinical trial protocols in the last twelve (12) months (CNS Resolution 251 of August 7, 1997, Part III, sub-item J), unless the investigator considers that there may be a direct benefit to the patient;
* Any observational finding (clinical/ physical evaluation), laboratory abnormality, disease or therapy that is interpreted by the investigator as a risk to the research participant's participation in the clinical trial;
* Aspartate transaminase (AST) or alanine aminotransferase (ALT) more than two times the normal upper limit of the central laboratory reference range after treatment with Simvastatin 20 mg for four weeks;
* Creatine phosphokinase (CPK) more than three times the normal upper limit of the central laboratory reference range after treatment with Simvastatin 20 mg for four weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Fonseca, physician, Principal Investigator — Universidade Federal de São Paulo
Locations (7):
- Brazil (7):
  - Centro de Pesquisas em Diabetes e Doenças Endócrino-Metabólicas- UFC, Fortaleza, Ceará
  - Centro de Pesquisas Médicas Básica e Clínica, Recife, Pernambuco
  - CCBR Brasil Centro de Pesquisas e Análises Clínicas, Rio de Janeiro
  - CEPIC Centro Paulista de Investigação Clínica, São Paulo
  - FGM - Clínica Paulista de Doenças Cardiovasculares, São Paulo
  - Hospital do Rim e Hipertensão, São Paulo
  - Universidade Federal de São Paulo, São Paulo

REFERENCES:
- [Derived] Vattimo ACA, Fonseca FAH, Morais DC, Generoso LF, Herrera R, Barbosa CM, de Oliveira Izar MC, Cardoso RA, Zung S. Efficacy and Tolerability of a Fixed-Dose Combination of Rosuvastatin and Ezetimibe Compared with a Fixed-Dose Combination of Simvastatin and Ezetimibe in Brazilian Patients with Primary Hypercholesterolemia or Mixed Dyslipidemia: A Multicenter, Randomized Trial. Curr Ther Res Clin Exp. 2020 Jul 28;93:100595. doi: 10.1016/j.curtheres.2020.100595. eCollection 2020. PMID 32904162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 7 research centers between March 2013 and July 2014. The first participant was enrolled on March 21, 2013 and the last participant was enrolled in July, 2014.
Pre-assignment Details: Of 637 recruited participants, 254 met eligibility criteria and were recruited in the run-in phase.The participants received Simvastatin 20 mg tablet orally once daily for 5 weeks in this period and 241 completed the run-in phase. Of the 241 participants, 129 were eligible for the treatment phase and randomized.
Period: Overall Study
Arm/Group | Rosuvastatin + Ezetimibe | Simvastatin + Ezetimibe
Started (Treatment (Open- label / 9 weeks)) | 66 | 63
Completed | 59 | 58
Not Completed | 7 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Non-adherence to medication | 4 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin + Ezetimibe | Simvastatin + Ezetimibe | Total
Number analyzed (Participants) | 66 | 63 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 41 | 90
  >=65 years | 17 | 22 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.39 (8.7) | 59.16 (9.6) | 59.28 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 53 | 108
  Male | 11 | 10 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 51 | 45 | 96
  More than one race | 9 | 12 | 21
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 66 | 63 | 129

OUTCOME MEASURES:

1. Primary Outcome: Reduction of LDL Cholesterol Levels
Description: The primary efficacy variable was the percentage of LDL-C variation at the end of nine weeks of treatment, compared to baseline (pre-randomization), in participants who achieved LDL <100 mg/dL were considered to have been successfully treated.
Time Frame: Baseline compared to the end of 9 weeks of treatment
Population: All randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change of LDL
Arm/Group | Rosuvastatin + Ezetimibe | Simvastatin + Ezetimibe
Number analyzed (Participants) | 66 | 63
percent change of LDL | -39.45 [-43.53 to -35.08] | -29.13 [-34.05 to -23.85]
Statistical Analysis 1: Comparison: Rosuvastatin + Ezetimibe vs Simvastatin + Ezetimibe; Rosuvastatin + Ezetimibe versus Simvastatin + Ezetimibe; Test type: Non-Inferiority — The non-inferiority assessment was analyzed by the bilateral confidence interval (95%) for the ratio of the mean LDLfinal/LDLbaseline of the R/E combination, compared to the mean LDLfinal/LDLbaseline of the S/E combination and the bilateral confidence interval (95%) for the difference between the two means of the percentage variation of LDL-C in the treatments ([(LDLfinal - LDLbaseline)/LDLbaseline))*100)R+E] - [(LDLfinal - LDLbaseline)/LDLbaseline))*100)S+E]; p = 0.0013, ANCOVA; Estimates for treatment effect and their 95% confidence intervals were exponentiated to produce estimates of percentage change; Median Difference (Final Values) = -10.32, 95% CI 2-sided [-16.94 to -3.70], Standard Error of Mean 3.33 — Mean Percentage Change LDL- C (%)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Rosuvastatin + Ezetimibe | Simvastatin + Ezetimibe
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/66 | 2/63
Other Adverse Events (participants affected / at risk) | 2/66 | 4/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin + Ezetimibe (N=66) | Simvastatin + Ezetimibe (N=63)
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pneumonia NOS (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin + Ezetimibe (N=66) | Simvastatin + Ezetimibe (N=63)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and the period of this evaluation is at least 45 days in advance. The sponsor can require changes to the communication or cannot approve it.